CLINICAL TRIAL: NCT05086887
Title: Infections in Migrants in Sweden - the Importance of Malaria and Other Parasitic Infections
Acronym: MMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: MMS2019
Record Dates: First submitted 2021-08-31; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Malaria; Parasitic Infection
Keywords: Migrant health; Malaria; Asymptomatic infections; Parasite prevalence; Screening
MeSH Terms: conditions — Malaria; Parasitic Diseases; Asymptomatic Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Peripheral blood 10ml, except in small children where 5ml are collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Migrants from malaria endemic countries arriving to or living in Sweden: The study population consists of participants born in a malaria endemic country living in Sweden, irrespective of time of residency in Sweden (e.g newly arrived migrants as well as individuals with longer residency in Sweden or another non-endemic country). Participants of all ages can be included in the study.
  Interventions: Diagnostic Test: Malaria diagnostic tests (RDT and PCR) and serology for malaria and other parasitic diseases

INTERVENTIONS:
Diagnostic Test: Malaria diagnostic tests (RDT and PCR) and serology for malaria and other parasitic diseases — All individuals are tested. Individuals with demonstrated parasitic disease are referred to the Infectious diseases or Pediatric clinic for evaluation and treatment.

SUMMARY:
Malaria is a parasitic disease causing substantial morbidity and mortality globally. Malaria is a potentially severe and fatal disease in non-immune individuals. In areas of intense transmission infections individuals acquired immunity that protect against clinical disease. Nonetheless, immunity is not regarding sterilizing and repeated infections often result in an asymptomatic carriage of malaria parasites. These chronic apparently asymptomatic infections have been associated with anemia, cognitive dysfunction and adverse events during pregnancy.

Global migration has increased over the last decade and has resulted in an increasing number of migrants from malaria endemic regions arriving in non-endemic countries. Migrants from malaria endemic countries may carry asymptomatic infections with malaria parasites, as well as other parasitic infections such as strongyloides and schistosomiasis, with a possible negative impact on health in this group. The prevalence of asymptomatic malaria and other parasites is not fully elucidated in migrants from different regions. Moreover, the longevity of asymptomatic carriage of malaria parasites in absence of re-exposure is not known.

The aim of this study is to assess the prevalence of malaria parasites and other parasitic infections in migrants in Sweden, both newly arrived and migrants with longer residency, and intend to evaluate the need for screening for various parasitic infections in migrants arriving in Sweden. Moreover, this study will also assess antibody responses to malaria and other parasitic diseases.

DETAILED DESCRIPTION:
Study participants are recruited in different ways, participation in the study is offered when attending an asylum health clinic at several sites in the Stockholm county. Secondly, patients attending the Infectious Disease outpatient clinic for non-febrile diseases (e.g. follow up of hepatitis, treatment for latent tuberculosis). Thirdly, quota refugees from Democratic Republic of the Congo or Uganda with arrival in Sweden in the years 2015-2019 with postal address in Stockholm, will be invited by letter to participate in the study .

A venous blood sample (EDTA tube) is collected from study participants at one occasion and a questionnaire including questions about patient origin and previous malaria are completed with the aid of a translator.

Blood samples are analysed in the research laboratory, where a malaria rapid diagnostic test (RDT) is performed and haemoglobin concentrations are measured (using Hemocue, point of care test) the same day as sample collection. The samples are then centrifuged, aliquoted, and stored frozen at the research laboratory. Presence of malaria parasites are analysed by realtime-PCR of the species specific 18SRNA gene in a multiplex assay. Serologic markers for other parasitic diseases (eg. schistosomiasis and strongyloides) are analysed in plasma. These analyses are performed at the reference laboratory at the Public Health Agency of Sweden.

Projected sample size is estimated using the formula n=(Z^2xP(1-P))/d^2 where P is the expected prevalence based on previous studies (5%) and d is the precision (1.5%) and Z is the confidence interval (95%). Based on these assumptions, the required sample size is n=715.

All RDT or PCR positive individuals are referred to the Department of Infectious Diseases or the Department of Pediatrics at the regional hospital for further investigations and treatment. Results from complete blood count are assessed and followed up according to clinical routine at each centre where samples were collected. Contact information to the study participant are included as part of the recruitment and consent procedures in order to be able to contact the study participants for referral.

Moreover, antibody responses to crude parasite extracts and specific antigens are assessed by ELISA and Luminex. In a subset of participants peripheral blood mononuclear cells, PBMC, are prepared in follow up samples to assess the cellular immune response. The magnitude and breadth of antibody and cellular responses are assessed in relation to duration of residency in a malaria free country. An estimation of the long- term decay kinetics using a sero-epidemiological mathematical model is performed.

All data will be handled according to the EU GDPR (General Data Protection Regulation) superseded all EU member states' data protection laws based on the 1995 Data Protection Directive (DPD), (GDPR, EU 2016/679 and SFS 2018:218). The patient register, containing all collected data and analysis results, is kept pseudonymizised and stored in a secure server at Karolinska University Hospital. The key to pseudonumization is kept in a secure locker at the institution.

Collected blood specimens are stored in Stockholm Medical Biobank located at Karolinska University Hospital in Solna. Handling of these stored samples is governed by the Act on Biobanks in Health Care (SFS 2002: 297).

ELIGIBILITY:
Inclusion Criteria:

* Born in a malaria endemic country (a country with reported indigenous spread of malaria according to World Malaria Report 2019)

Exclusion Criteria:

* Inability to understand study information or sign informed consent, except for children where legal guardian is asked for consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Migrants born in countries where malaria is endemic are invited to participate in the study at migration health care units and in the antenatal care during pregnancy.
  2. Immigrants from malaria endemic countries living in Sweden are invited to participate with voluntary blood sampling on one occasion. The study is advertised in posters in waiting areas at health clinics.
  3. Family members to individuals that are diagnosed with malaria at Karolinska University Hospital or other hospitals in Stockholm and Västerås are invited to the study at in-patient clinics.
  4. Persons with origin in Democratic Republic of the Congo and Uganda arrived in Sweden between 2015-2019 are invited by an addressed letter
Sampling Method: Non-Probability Sample
Enrollment: 715 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Parasite prevalence | Measured at one occasion within 10 years from arrival in Sweden
  Number of participants with ongoing malaria infection
Prevalence of other parasites focusing on strongyloides and schistosomiasis | Measured at one occasion within 10 years from arrival in Sweden
  Number of participants showing serological response to strongyloides and schistosomiasis

SECONDARY OUTCOMES:
Immune responses to malaria and other parasites | A blood specimen will be collected from participants upon inclusion, and a subset of volunteers will be asked to contribute with a second blood sample after 6-12 months
  Levels and breadth of P. falciparum specific antibody and memory B cell responses.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Farnert, MD, Prof, Principal Investigator — Karolinska University Hospital
Locations (1):
- Asylum Health Care Facilities in SLSO and Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] White NJ, Pukrittayakamee S, Hien TT, Faiz MA, Mokuolu OA, Dondorp AM. Malaria. Lancet. 2014 Feb 22;383(9918):723-35. doi: 10.1016/S0140-6736(13)60024-0. Epub 2013 Aug 15. PMID 23953767
- [Background] Doolan DL, Dobano C, Baird JK. Acquired immunity to malaria. Clin Microbiol Rev. 2009 Jan;22(1):13-36, Table of Contents. doi: 10.1128/CMR.00025-08. PMID 19136431
- [Background] Babiker HA, Abdel-Muhsin AM, Ranford-Cartwright LC, Satti G, Walliker D. Characteristics of Plasmodium falciparum parasites that survive the lengthy dry season in eastern Sudan where malaria transmission is markedly seasonal. Am J Trop Med Hyg. 1998 Oct;59(4):582-90. doi: 10.4269/ajtmh.1998.59.582. PMID 9790434
- [Background] Sifft KC, Geus D, Mukampunga C, Mugisha JC, Habarugira F, Fraundorfer K, Bayingana C, Ndoli J, Umulisa I, Karema C, von Samson-Himmelstjerna G, Aebischer T, Martus P, Sendegeya A, Gahutu JB, Mockenhaupt FP. Asymptomatic only at first sight: malaria infection among schoolchildren in highland Rwanda. Malar J. 2016 Nov 14;15(1):553. doi: 10.1186/s12936-016-1606-x. PMID 27842542
- [Background] Fernando SD, Rodrigo C, Rajapakse S. The 'hidden' burden of malaria: cognitive impairment following infection. Malar J. 2010 Dec 20;9:366. doi: 10.1186/1475-2875-9-366. PMID 21171998
- [Background] Okell LC, Bousema T, Griffin JT, Ouedraogo AL, Ghani AC, Drakeley CJ. Factors determining the occurrence of submicroscopic malaria infections and their relevance for control. Nat Commun. 2012;3:1237. doi: 10.1038/ncomms2241. PMID 23212366
- [Background] Asghar M, Hasselquist D, Hansson B, Zehtindjiev P, Westerdahl H, Bensch S. Chronic infection. Hidden costs of infection: chronic malaria accelerates telomere degradation and senescence in wild birds. Science. 2015 Jan 23;347(6220):436-8. doi: 10.1126/science.1261121. PMID 25613889
- [Background] Marangi M, Di Tullio R, Mens PF, Martinelli D, Fazio V, Angarano G, Schallig HD, Giangaspero A, Scotto G. Prevalence of Plasmodium spp. in malaria asymptomatic African migrants assessed by nucleic acid sequence based amplification. Malar J. 2009 Jan 12;8:12. doi: 10.1186/1475-2875-8-12. PMID 19138412
- [Background] Matisz CE, Naidu P, Shokoples SE, Grice D, Krinke V, Brown SZ, Kowalewska-Grochowska K, Houston S, Yanow SK. Post-arrival screening for malaria in asymptomatic refugees using real-time PCR. Am J Trop Med Hyg. 2011 Jan;84(1):161-5. doi: 10.4269/ajtmh.2011.10-0494. PMID 21212221
- [Background] Maroushek SR, Aguilar EF, Stauffer W, Abd-Alla MD. Malaria among refugee children at arrival in the United States. Pediatr Infect Dis J. 2005 May;24(5):450-2. doi: 10.1097/01.inf.0000160948.22407.0d. PMID 15876946
- [Background] Monge-Maillo B, Lopez-Velez R. Migration and malaria in europe. Mediterr J Hematol Infect Dis. 2012;4(1):e2012014. doi: 10.4084/MJHID.2012.014. Epub 2012 Mar 10. PMID 22536477
- [Background] Karki T, Napoli C, Riccardo F, Fabiani M, Dente MG, Carballo M, Noori T, Declich S. Screening for infectious diseases among newly arrived migrants in EU/EEA countries--varying practices but consensus on the utility of screening. Int J Environ Res Public Health. 2014 Oct 21;11(10):11004-14. doi: 10.3390/ijerph111011004. PMID 25337945
- [Background] Monge-Maillo B, Lopez-Velez R. Is screening for malaria necessary among asymptomatic refugees and immigrants coming from endemic countries? Expert Rev Anti Infect Ther. 2011 May;9(5):521-4. doi: 10.1586/eri.11.37. PMID 21609263
- [Background] Chaves NJ, Paxton GA, Biggs BA, Thambiran A, Gardiner J, Williams J, Smith MM, Davis JS. The Australasian Society for Infectious Diseases and Refugee Health Network of Australia recommendations for health assessment for people from refugee-like backgrounds: an abridged outline. Med J Aust. 2017 Apr 17;206(7):310-315. doi: 10.5694/mja16.00826. PMID 28403765
- [Background] Stauffer WM, Weinberg M, Newman RD, Causer LM, Hamel MJ, Slutsker L, Cetron MS. Pre-departure and post-arrival management of P. falciparum malaria in refugees relocating from sub-Saharan Africa to the United States. Am J Trop Med Hyg. 2008 Aug;79(2):141-6. PMID 18689612
- [Background] Njama-Meya D, Kamya MR, Dorsey G. Asymptomatic parasitaemia as a risk factor for symptomatic malaria in a cohort of Ugandan children. Trop Med Int Health. 2004 Aug;9(8):862-8. doi: 10.1111/j.1365-3156.2004.01277.x. PMID 15303990
- [Background] Szmitko PE, Kohn ML, Simor AE. Plasmodium falciparum malaria occurring 8 years after leaving an endemic area. Diagn Microbiol Infect Dis. 2009 Jan;63(1):105-7. doi: 10.1016/j.diagmicrobio.2008.08.017. Epub 2008 Oct 21. PMID 18945569
- [Background] Cowman AF, Healer J, Marapana D, Marsh K. Malaria: Biology and Disease. Cell. 2016 Oct 20;167(3):610-624. doi: 10.1016/j.cell.2016.07.055. PMID 27768886
- [Background] Langhorne J, Ndungu FM, Sponaas AM, Marsh K. Immunity to malaria: more questions than answers. Nat Immunol. 2008 Jul;9(7):725-32. doi: 10.1038/ni.f.205. PMID 18563083
- [Background] Farnert A, Wyss K, Dashti S, Naucler P. Duration of residency in a non-endemic area and risk of severe malaria in African immigrants. Clin Microbiol Infect. 2015 May;21(5):494-501. doi: 10.1016/j.cmi.2014.12.011. Epub 2014 Dec 26. PMID 25656623
- [Background] Shokoples SE, Ndao M, Kowalewska-Grochowska K, Yanow SK. Multiplexed real-time PCR assay for discrimination of Plasmodium species with improved sensitivity for mixed infections. J Clin Microbiol. 2009 Apr;47(4):975-80. doi: 10.1128/JCM.01858-08. Epub 2009 Feb 25. PMID 19244467
- [Background] Rono J, Osier FH, Olsson D, Montgomery S, Mhoja L, Rooth I, Marsh K, Farnert A. Breadth of anti-merozoite antibody responses is associated with the genetic diversity of asymptomatic Plasmodium falciparum infections and protection against clinical malaria. Clin Infect Dis. 2013 Nov;57(10):1409-16. doi: 10.1093/cid/cit556. Epub 2013 Aug 27. PMID 23983244
- [Background] Yman V, White MT, Rono J, Arca B, Osier FH, Troye-Blomberg M, Bostrom S, Ronca R, Rooth I, Farnert A. Antibody acquisition models: A new tool for serological surveillance of malaria transmission intensity. Sci Rep. 2016 Feb 5;6:19472. doi: 10.1038/srep19472. PMID 26846726

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05086887/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT05086887/ICF_001.pdf